CLINICAL TRIAL: NCT03431649
Title: Efficacy of Beraprost in Lowering Pulmonary Arterial Pressure in Pulmonary Arterial Hypertension Children Associated With Left to Right Shunt Congenital Heart Defect
Brief Title: Efficacy of Beraprost in Lowering Pulmonary Arterial Pressure in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Soetomo General Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. dr. Mahrus A. Rahman Sp.A(K), Doctor, Dr. Soetomo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAshirley
Record Dates: First submitted 2017-07-29; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Pediatric Pulmonary Hypertension
MeSH Terms: interventions — beraprost; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: the researchers don't know which drug taken by the patient and don't know the previous PA pressure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Beraprost Sodium (Experimental): Beraprost 1mcg/kg/day, divided in 3 doses orally patient was followed up for 12 weeks, then echocardiography evaluation was performed in patient completed the study.
  22 patients
  Interventions: Drug: Beraprost Sodium
- Sildenafil citrate (Active Comparator): Sildenafil 0.4 mg/kg/time, 4 times daily per oral patient was followed up for 12 weeks, then echocardiography evaluation was performed in patient completed the study.
  20 patients
  Interventions: Drug: Sildenafil Citrate

INTERVENTIONS:
Drug: Beraprost Sodium — 1 mcg /kgbw daily, divided in three dosages orally for 12 weeks
  Other Names: Dorner
  Arms: Beraprost Sodium
Drug: Sildenafil Citrate — 0.4 mg/kgbw each time, 4 times in a day orally for 12 weeks
  Other Names: Viagra
  Arms: Sildenafil citrate

SUMMARY:
To analyze the efficacy of beraprost and sildenafil for treatment of pulmonary hypertension in children with left to right shunt.

analyze the efficacy and side effects.

DETAILED DESCRIPTION:
Eligibility criteria:

Inclusion:

1. children aged 1-17 years with left to right shunt, diagnosed as pulmonary hypertension.
2. free from chronic pulmonary disease
3. never performed any cardiac surgical
4. never got any treatment for PH
5. agree to enroll in this study. Exclusion

1. suffer from portal hypertension, HIV and connective tissue disease 2. under interferon therapy.

Outcome measure:

Pulmonary artery pressure

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as pulmonary hypertension with left to right shunt CHD (VSD, ASD, PDA and combination)
* agree to enroll in this study

Exclusion Criteria:

* suffer from chronic lung disease
* suffer from soft tissue tumor, HIV/AIDS
* under interferon therapy
* already performed any cardiac surgery
* already got anti-PH remedy

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of Beraprost, Sildenafil and comparison between both drugs in lowering pulmonary arterial pressure | 12 weeks
  Measuring mPAP (pre-post therapy) via echocardiography before and after consuming sildenafil or beraprost

SECONDARY OUTCOMES:
Emergent Adverse Events | 12 weeks
  adverse event reported by patients and during weekly examination after consuming Beraprost or Sildenafil: hypotension, dizzy, headache, flushing, bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Mahrus Rachman, MD, Study Director — Dr. Soetomo General Hospital
Locations (1):
- Dr. Soetomo General Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Limsuwan A, Pienvichit P, Khowsathit P. Beraprost therapy in children with pulmonary hypertension secondary to congenital heart disease. Pediatr Cardiol. 2005 Nov-Dec;26(6):787-91. doi: 10.1007/s00246-005-0925-4. PMID 16132278